CLINICAL TRIAL: NCT04636632
Title: Weekly Fosaprepitant for the Prevention of Nausea and Emesis During Concurrent Chemoradiotherapy for Nasopharyngeal Carcinoma: a Prospective Pilot Study
Brief Title: Fosaprepitant for the Prevention of Nausea and Emesis During Concurrent Chemoradiotherapy for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSUCC-MYC-2020-1104
Record Dates: First submitted 2020-11-10; First posted 2020-11-19 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — fosaprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Arm (Experimental): fosaprepitant 150mg/m2 weekly in concurrent with radiotherapy during concurrent chemoradiotherapy
  Interventions: Drug: fosaprepitant
- Triweekly Arm (Active Comparator): fosaprepitant 150mg/m2 triweekly in concurrent with chemotherapy during concurrent chemoradiotherapy
  Interventions: Drug: fosaprepitant

INTERVENTIONS:
Drug: fosaprepitant — fosaprepitant 150mg/m2 weekly or triweekly during concurrent chemoradiotherapy

SUMMARY:
This is an opene-label, single center, randomized prospective pilot study to compare the efficacy of weekly versus triweekly fosaprepitant regimens for the prevention of nausea and emesis during concurrent chemoradiotherapy for nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
Scheme:

Eligible fosaprepitant sensitive (complete response [defined as no emesis and no use of rescue antiemetics] during the overall phase [0 to 120 hours] of all cycles of cisplatin-based induction chemotherapy) NPC patients will be randomized to 2 arms at 1:1 ratio.

* Weekly Arm: fosaprepitant 150mg/m2 weekly in concurrent with radiotherapy during concurrent chemoradiotherapy.
* Triweekly Arm: fosaprepitant 150mg/m2 triweekly in concurrent with chemotherapy during concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* Stage II - IVa NPC patients (according to the 8th AJCC edition)
* Male and no pregnant female
* Scheduled for cisplatin-based induction chemotherapy (cisplatin≥ 70 mg/m2)and concomitant triweekly cisplatin
* Fosaprepitant sensitive (complete response [defined as no emesis and no use of rescue antiemetics] during the overall phase [0 to 120 hours] of all cycles of cisplatin-based induction chemotherapy)
* Age between 18-70
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <2.0×upper limit of normal (ULN)
* Adequate renal function: creatinine clearance ≥60 ml/min
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70
* Without radiotherapy or chemotherapy
* Patients must give signed informed consent

Exclusion Criteria:

* Evidence of relapse or distant metastasis
* Pregnancy or lactation
* History of prior malignancy or previous treatment for NPC
* Had other current malignant diagnoses apart from non-melanoma skin cancers
* Emesis or clinically significant nausea (moderate or severe) in the 24 h before the first dose of study medication
* Drugs with antiemetic activity were not allowed for the 24 h before receiving the first dose of study medication
* Known history of central nervous system disease (e.g., a seizure disorder or brain metastases )
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
the proportion of subjects with complete response (CR) overall | 7 weeks
  defined as no emesis and no use of rescue therapy

SECONDARY OUTCOMES:
the proportion of subjects with complete control (CC) overall | 7 weeks
  defined as no emesis and no use of rescue therapy and no significant nausea
the proportion of subjects with sustained no emesis overall | 7 weeks
the proportion of subjects with no nausea overall | 7 weeks
the proportion of subjects with no significant nausea overall | 7 weeks
  defined as no or mild nausea
the proportion of subjects with CR in the 24 hours following initiation of radiotherapy and concomitant cisplatin | 24 hours
  defined as no emesis and no use of rescue therapy
the proportion of subjects with CR in the 120 hours following initiation of radiotherapy and concomitant cisplatin | 120 hours
  defined as no emesis and no use of rescue therapy
the mean time to first emetic episode | 7 weeks
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) overall | 7 weeks
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) overall | 7 weeks

OTHER OUTCOMES:
Progress-free survival (PFS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yang Q, Zou X, Xie YL, Lin C, Ouyang YF, Liu YL, Duan CY, You R, Liu YP, Liu RZ, Huang PY, Guo L, Hua YJ, Chen MY. Fosaprepitant Weekly vs Every 3 Weeks for the Prevention of Concurrent Chemoradiotherapy-Induced Nausea and Vomiting: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2326127. doi: 10.1001/jamanetworkopen.2023.26127. PMID 37498596